CLINICAL TRIAL: NCT00792116
Title: The Effects of Gum Chewing on Standardized Math Scores in Adolescents
Brief Title: The Effects of Gum Chewing on Math Scores in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Children's Nutrition Research Center (Other)
Responsible Party: Craig Johnston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: gum and math scores
Record Dates: First submitted 2008-10-24; First posted 2008-11-17 (Estimated); Results first posted 2008-11-17 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Academic Achievement in Math
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Gum Chewing (Experimental)
  Interventions: Behavioral: Gum Chewing
- Non-gum chewing (No Intervention)

INTERVENTIONS:
Behavioral: Gum Chewing
  Arms: Gum Chewing

SUMMARY:
Context: Gum chewing has been shown to increase cognitive functioning. With the rise in standardized testing of school-age children and the concurrent attempts to improve their scores, finding simple and inexpensive methods to bolster performance is needed.

Objective: To examine the effects of gum chewing on standardized test scores and class grades in a group of 8th grade math students.

Design: Math classes were randomized to a gum chewing (GC) condition that provided students with gum during class and testing, or a control condition with no gum (NG) provided during class and testing. This study was conducted during the Spring 2008 school semester.

Setting: A charter school in Houston, TX.

Participants: All students enrolled in eighth grade math at the charter school were approached for recruitment in this study. A total of 108 (94%) students participated. Participants were between the ages of 13 and 16.

Main Outcome Measures: The Texas Assessment of Knowledge and Skills (TAKS), the Woodcock Johnson III Tests of Achievement (WJ-III), and math class grades were used to assess any differences in academic performance between the GC and NGC conditions. For purposes of this study, only the math sections of the WJ-III and TAKS, which are both standardized tests, were assessed.

Our primary hypothesis was that adolescents in a gum chewing (GC) condition would have significantly improved standardized test scores and math grades compared to adolescents in a non-gum chewing (NG) control condition.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in eight grade math class

Exclusion Criteria:

* Parents did not consent to participation

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

REFERENCES:
- [Derived] Johnston CA, Tyler C, Stansberry SA, Moreno JP, Foreyt JP. Brief report: gum chewing affects standardized math scores in adolescents. J Adolesc. 2012 Apr;35(2):455-9. doi: 10.1016/j.adolescence.2011.04.003. Epub 2011 May 26. PMID 21620465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Researchers and school personnel contacted the parents of all students (n=115) enrolled in an eighth grade math class during the Spring 2008 semester at a charter school in Houston, TX to participate in the current study. A total of 108 (94%) parents provided consent for their children to participate in the study.
Period: Overall Study
Arm/Group | Gum Chewing | Non-Gum Chewing
Started | 53 | 55
Completed | 52 | 54
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Discontnued intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gum Chewing | Non-Gum Chewing | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 55 | 108
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.7 (.8) | 14.6 (.7) | 14.6 (.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Math Scores on the Texas Assessment of Knowledge and Skills (TAKS)
Description: The TAKS test is a statewide standardized test administered to all Texas schoolchildren (15). The TAKS assesses reading, math, science, and social studies for 8th grade students; however, the current study analyzed only math scores.
Time Frame: the beginning of a school semester
Population: 106 participants were analyzed. One particiapant relocated to another school and one participant was removed by the teacher for discipline reasons.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Gum Chewing | Non-Gum Chewing
Number analyzed (Participants) | 52 | 54
percentile | 65.1 (14.0) | 70.0 (14.16)

2. Primary Outcome: Math Grades
Time Frame: baseline (the beginning of a school semester )
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average percentage correct
Arm/Group | Gum Chewing | Non-Gum Chewing
Number analyzed (Participants) | 52 | 54
average percentage correct | 77.7 (8.4) | 80.8 (7.63)

3. Secondary Outcome: Math Scores on the Woodcock Johnson III Tests of Achievement (WJ-III)
Description: The WJ-III (10) is a standardized test battery used to assess an individual's academic strengths and weaknesses. For purposes of the current study, students were given the 4 math subtests of the WJ-III.
Time Frame: the beginning of a school semester and 14 weeks later (the end of a school semester)
Reporting Status: Not Posted
Measure: Number (Standard Deviation)

4. Secondary Outcome: Scores on the Math Anxiety Rating Scale for Adolescents (MARS-A)
Description: he MARS-A (12) is a 98-item scale that lists various everyday situations in which adolescents may have to use mathematics.
Time Frame: the beginning of a school semester and 14 weeks later (the end of a school semester)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation)

5. Secondary Outcome: State Anxiety Scores on the State Trait Anxiety Index for Children (STAIC).
Description: The STAIC is a scale that distinguishes between a situationally based anxiety and a general intrinsic inclination towards experiencing feelings of anxiety
Time Frame: the beginning of a school semester and 14 weeks later (the end of a school semester)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation)

6. Primary Outcome: Math Scores on the Texas Assessment of Knowledge and Skills (TAKS).
Description: as for outcome 1
Time Frame: 14 weeks (end of the semester)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Gum Chewing | Non-Gum Chewing
Number analyzed (Participants) | 52 | 54
percentile | 84.9 (10.3) | 85.7 (11.4)
Statistical Analysis 1: Comparison: Gum Chewing vs Non-Gum Chewing; Test type: Non-Inferiority or Equivalence; p = .05, ANCOVA; Repeated Measures

7. Primary Outcome: Math Grades
Time Frame: 14 week (end of the semester)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average percentage correct
Arm/Group | Gum Chewing | Non-Gum Chewing
Number analyzed (Participants) | 52 | 54
average percentage correct | 75.2 (8.4) | 76.40 (8.8)
Statistical Analysis 1: Comparison: Gum Chewing vs Non-Gum Chewing; Test type: Non-Inferiority or Equivalence; p = .05, ANCOVA; Repeated Measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes